CLINICAL TRIAL: NCT06535672
Title: The Effect of Diabetes Education Given to Children Diagnosed With Type 1 Diabetes Mellitus Using the Kamishibai Method on Patients' Knowledge Level, HbA1c Parameter, and Quality of Life: A Randomized Controlled Trial
Brief Title: The Effect of Kamishibai Diabetes Education on Knowledge, HbA1c, and Quality of Life in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Makbule Yelda KARADERE REZAEE, Diabetes Training Nurse, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/99
Record Dates: First submitted 2024-06-13; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: DIABETES EDUCATION
Keywords: Type 1 Diabetes Mellitus (Type 1 DM); Kamishibai method; Hemoglobin A1c (HbA1c); Pediatric diabetes education; Quality of life in children; Randomized controlled tria
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Stratified randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kamishibai Diabetes Education (Experimental): Patients in the intervention group will receive diabetes education using the Kamishibai method. This method involves interactive storytelling tailored to the cognitive and sensory development of children aged 8-12. Training will be conducted over 3 days, with 3 sessions each day.
  Patients will attend training daily without hospitalization. Training includes interactive storytelling using the Kamishibai method, designed to be engaging and suitable for children aged 8-12.
  After the training, participants will complete the Diabetes Knowledge Level Evaluation Form, the PedsQL 3.0 Quality of Life Scale, and the Kamishibai Training Feedback Form. Filling out the forms will take approximately 30 minutes.
  Follow-up information and checks will be provided every 3 months.
  Interventions: Other: kamishibai education
- Routine diabetes education (Experimental): Patients in the control group will receive routine diabetes education as per standard hospital procedures. This training will also occur over 3 days, with 3 sessions per day.
  Training involves a PowerPoint presentation and a whiteboard, based on the Ministry of Health Childhood Diabetes Education guide.
  The language used will be simple and understandable for children. The training will be interactive, encouraging feedback and questions. Participants will fill out the Diabetes Knowledge Level Evaluation Form, PedsQL 3.0 Quality of Life Scale, and Routine Education Feedback Form after the training.
  Filling out the forms will take approximately 30 minutes. Follow-up information and checks will be provided every 3 months.
  Interventions: Other: routine education

INTERVENTIONS:
Other: kamishibai education — Patients in the intervention group will be given Kamishibai diabetes education.
  Arms: Kamishibai Diabetes Education
Other: routine education — Patients in the control group will be given routine diabetes education.
  Other Names: Patients in the intervention group will be given Kamishibai diabetes education.
  Arms: Routine diabetes education

SUMMARY:
Children diagnosed with Type 1 Diabetes Mellitus (T1DM) initially receive intensive education with their families. Studies indicate that over time, this initial education becomes routine, reducing its effectiveness and failing to adequately address developmental stages, thus requiring repetition. Current methods involve long and intensive educational sessions in hospitals using the Childhood Diabetes Education Guide. These extended, non-interactive sessions often lead to a loss of motivation, decreased learning efficiency, and negative attitudes among patients and their families.

This study aims to develop an educational tool utilizing the Kamishibai method specifically for children with T1DM aged 8-12. The Kamishibai method is designed to align with their cognitive and sensory development, promoting effective and engaging learning experiences for diabetic patients. By incorporating interactive and visually stimulating elements, Kamishibai seeks to enhance motivation and retention of diabetes education.

Hypothesis 1: Children diagnosed with Type 1 DM have higher knowledge levels in the group educated with the Kamishibai method compared to those receiving routine education.

Hypothesis 2: The Hemoglobin A1c parameter is lower in the Kamishibai-educated group.

Hypothesis 3: The quality of life is higher in the Kamishibai-educated group.

This study will assess the effectiveness of the Kamishibai method by comparing it to routine educational approaches. The detailed protocol includes technical aspects of the intervention, measurement tools, data collection methods, and statistical analysis plans to ensure a comprehensive evaluation of the method's impact on knowledge levels, HbA1c parameters, and quality of life.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to examine the impact of diabetes education using the Kamishibai method on knowledge levels, HbA1c parameters, and quality of life in children diagnosed with T1DM. The study protocol is detailed below.

Data Collection Tools: The Child Information Form, Diabetes Knowledge Level Evaluation Form, PedsQL 3.0 Quality of Life Scale for Children with Type 1 Diabetes (Child Form), Blood Sugar and HbA1c Monitoring Diary, and Kamishibai Education Feedback Form will be used.

Implementation:

The study data will be collected using a stratified random sampling method. Children aged 8-12 years who meet the inclusion criteria will be stratified by their HbA1c values and divided into two groups by block randomization (n=30 intervention, n=30 control). The intervention group will receive Kamishibai diabetes education, while the control group will receive routine diabetes education. Information about the study will be provided to eligible children and parents. Informed consent will be obtained from those agreeing to participate. Data collection forms will be filled out. Each child will have follow-up diabetes nurse appointments 1 week after the education and doctor appointments 10 days later.

Intervention Group (n=30):

Patients in the intervention group will receive Kamishibai diabetes education, completed over 3 days with 3 sessions per day. Post-education data collection forms will be administered, taking approximately 30 minutes to complete. Patients will be informed about follow-up checks and the process for the next 3 months.

Control Group (n=30):

Patients in the control group will receive routine diabetes education over 3 days with 3 sessions per day. The education will use a PowerPoint presentation and a whiteboard according to the Ministry of Health's Childhood Diabetes Education guide. Simple, understandable language will be used for children's comprehension. The education will be interactive, encouraging feedback and questions.

Form and Metabolic Tests Application at the 3rd and 6th Month:

At the 3rd and 6th months post-education, patients attending doctor check-ups will visit the diabetes education unit. HbA1c and data collection forms will be administered 3 and 6 months post-education. Filling out the forms will take approximately 15-20 minutes.

Population and Sample of the Study:

The study population consists of children aged 8-12 years (N=101) followed at Istanbul Zeynep Kâmil Women and Children's Diseases Training and Research Hospital between January 1, 2024, and April 29, 2024. The sample includes patients diagnosed with Type 1 Diabetes who meet the inclusion criteria from the population.

Inclusion Criteria for the Sample:

Children aged 8-12 years Being followed up for at least 1 year with a diagnosis of Type 1 diabetes Being followed as outpatients Using insulin Able to understand and speak Turkish

Exclusion Criteria for the Sample:

Presence of another chronic disease that could affect glycemic control apart from Type 1 diabetes Using an insulin pump Having vision and/or hearing problems Having mental and/or neurological issues Having a diagnosis of a psychiatric disorder

Exclusion Criteria from the Sample:

The child and/or family not wishing to continue the study The child not participating in the entire education program Diagnosis of a different disease affecting glycemic control during the study The child's treatment continuing in another institution Not attending the regular 3-month check-ups Dependent Variables: Patients' diabetes knowledge score, HbA1c values, and Quality of Life Scale score in children with Type 1 Diabetes.

Independent Variables: Diabetes education using the Kamishibai method, routine diabetes education.

Sample Size: Determined using G. POWER 3.1.9.7 (Heinrich-Heine-Universität Düsseldorf, Germany). Values from a study by Alzawahreh and Öztürk (2024) on adolescents diagnosed with T1DM were used for HbA1c scores. With a 5% alpha error (α=0.05), 10% beta error (β=0.10), and 0.80 power (d=0.804), a total of 60 participants (30 in the intervention group, 30 in the control group) were determined. Considering potential losses, the sample size was increased by 10%. The study is planned with 66 children (33 in the intervention group, 33 in the control group).

Data Collection: Written permission was obtained from the Ethics Committee of Zeynep Kamil Women and Children's Diseases Training and Research Hospital and research permission from the Istanbul Governorship Provincial Health Directorate. After explanations to families of eligible children, verbal and written informed consent will be obtained from participants' families. Personal information will be kept confidential, and their privacy will be respected during the study. Data will be collected between July 2024 and July 2025.

Data Analysis: The data will be analyzed using SPSS 26.0 (Statistical Package for Social Science). Arithmetic mean (Mean), standard deviation (SD), minimum and maximum values will be used for continuous variables. Frequency and percentage calculations will be used for categorical variables. Cronbach's alpha coefficient will determine the internal consistency of the scale items. The Kolmogorov-Smirnov test will assess normal data distribution. Non-parametric tests will be used if data do not show normal distribution. "Chi-square" and "Fisher exact" tests will compare groups with categorical data. The "Mann Whitney U" test will compare numerical data between groups and examine differences between scale averages. The "Friedman test" will examine numerical variable differences at different times within a group. "Spearman correlation" analysis will examine the relationship between scales. In all tests, p < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* The child is 8-12 years old.
* Diagnosed with Type 1 Diabetes Mellitus (T1DM) for at least 1 year.
* Followed up on an outpatient basis.
* The child is using insulin.
* The child can understand and speak Turkish.

Exclusion Criteria:

* Presence of another chronic disease other than T1DM that may affect glycemic control.
* Using an insulin pump.
* Having vision and/or hearing problems.
* Having a mental and/or neurological problem.
* Having a diagnosis of a psychiatric disease.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Assessed by the PedsQL 3.0 Child Form | At baseline, three months later, six months later (15 minutes ago)
  The PedsQL™ 3.0 Diabetes Module, developed by Varni et al. (2003), measures diabetes-specific quality of life in children. The Turkish validity study of this scale was conducted by Ayar and Öztürk (2016). The scale, consisting of a total of 28 items, includes five sub-dimensions:
  Diabetes-Related Problems (11 items) Treatment Barriers (4 items) Adherence to Treatment (7 items) Worry (3 items) Communication (3 items)
  The 5-point Likert scale is scored as follows:
  0 = Never
  1. = Rarely
  2. = Sometimes
  3. = Often
  4. = Always The total score ranges from 0 to 100. As the total score increases, the quality of life also increases. A score of 0 indicates never a problem (100 points), 1 indicates rarely a problem (75 points), 2 indicates sometimes a problem (50 points), 3 indicates often a problem (25 points), and 4 indicates always a problem (0 points).
HbA1c Value Assessed by Blood Test Results | At baseline, three months later, six months later (15 minutes ago)
  HbA1c is a glycosylated hemoglobin test that provides an average level of blood glucose over a 2-3 month period, indicating the average blood glucose values.
Diabetes Knowledge Level Assessed by the Diabetes Knowledge Level Evaluation Form | At baseline (5 minutes ago)
  The Diabetes Knowledge Level Evaluation Form is prepared by the researchers based on literature. The form consists of 20 questions covering the following areas:
  What is diabetes and how is it managed? (Questions 1-3) Insulin and blood sugar control (Question 4) Healthy eating (Questions 5-7) Exercise (Questions 8-10) Management of hyperglycemia and hypoglycemia (Questions 11-13) Diabetes management during illness (Questions 14-16) Diabetes management at school (Questions 17-18) General health and care (Question 19) Prevention of chronic complications (Question 20) Responses can be marked as correct, incorrect, or left blank. Correct answers are scored 1 point, while blank or incorrect answers are scored 0 points. The total knowledge score is calculated out of 20 points.

CONTACTS AND LOCATIONS:
Overall Officials: Gülzade Uysal, Assoc.Dr., Principal Investigator — Sakarya University of Applied Sciences Faculty of Health Sciences
Locations (1):
- Work, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No